CLINICAL TRIAL: NCT05934760
Title: Assessing the Impact of Age, and a Short-term High-intensity Interval Training (HIIT) on Skeletal Muscle Mass and Mitochondrial Activity
Acronym: Mi-HIIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Mi-HIIT CMMP
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Aging; Sarcopenia
Keywords: Exercise; Mitochondrial function; Healthy Aging
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Masking Description: Due to the nature of exercise interventions, it is not possible to blind the participants or investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (HIIT) (Experimental): Older participants (over 60) will be randomized to perform home-based unsupervised exercise, the HIIT group will perform the HIIT intervention 3 times a week, at home, unsupervised for 4 weeks. This will be supported by regular contact from a member of the research team to provide support and to encourage adherance.
  Our research group has conducted many similar exercise regimes of this intensity to subjects in the anticipated age-range without incident. Participants will be adviced to terminate exercise training immediately if experiencing:
  * Chest pain or tightness
  * Faintness
  * Sudden pallor
  * Loss of co-ordination
  * Confusion
  * Dizziness
  * Palpitations
  * Sudden breathlessness
  Should any participant experience these effects during any session, they will be advised to seek urgent medical attention and will be withdrawn from the exercise arm of the study for safety purposes.
  Interventions: Other: High intensity interval training (HIIT)
- Resistance exercise training (RET) (Experimental): Older participants (over 60) will be randomized to perform home-based unsupervised exercise, the RET group will perform the RET intervention at home, 3 times a week unsupervised for 4 weeks.This will be supported by regular contact from a member of the research team to provide support and to encourage adherance.
  Our research group has conducted many similar exercise regimes of this intensity to subjects in the anticipated age-range without incident. Participants will be adviced to terminate exercise training immediately if experiencing:
  * Chest pain or tightness
  * Faintness
  * Sudden pallor
  * Loss of co-ordination
  * Confusion
  * Dizziness
  * Palpitations
  * Sudden breathlessness
  Should any participant experience these effects during any session, they will be advised to seek urgent medical attention and will be withdrawn from the exercise arm of the study for safety purposes.
  Interventions: Other: Resistance based training (RET)

INTERVENTIONS:
Other: High intensity interval training (HIIT) — Each HIIT session last 15 minutes. Participants will be asked to measure their own heart rate during their rest periods and provided with an estimated max heart rate which they should be aiming to achieve within the final 2 exercises. Participants will be provided with a logbook to record the heart rate achieved in each exercise. The regimen will include:
  * 2 min warm-up: jogging on the spot
  * Each of the following exercises performed for 60seconds, interspaced by 90 seconds rest
    * Star jumps
    * Standing squats
    * On-the-spot sprints
    * Standing squats
    * Star jumps
  * 2 min cool-down: jogging on the spot
  Arms: High intensity interval training (HIIT)
Other: Resistance based training (RET) — Each RET session lasts an estimated 20minutes. Participants will be provided with a set of resistance bands to provide resistance to their workout, and a logbook to record the number of repetitions and band used.
  Each session will include:
  * 2 min warm-up jogging on the spot
  * 2 sets of 12-15 repetitions of:
  * Squats
  * Hip flexion
  * Hip extension
  * Hip abduction
  * Seated row
  * Bench press
  * Lateral raises
  * 2 min jogging on the spot cooldown.
  Each exercise will be separated by 1-minute rest, with participants encouraged to workout to mild fatigue on their final repetition in each set. If able to perform more than the allocated maximum of 15 repetitions prior to fatigue, then participants will be informed to increase the resistance by using a tougher resistance band.
  Arms: Resistance exercise training (RET)

SUMMARY:
The goal of this interventional study is to learn about the role of mitochondrial function in healthy aging, and then go on and assess the role of a home-based exercise program on the changes seen. The main question[s] it aims to answer are:

* What alterations in skeletal muscle mitochondrial function are seen in healthy aging?
* Can a short-term exercise program alter these alterations seen?

The older participants will be invited to take part in a home-based 4 week exercise intervention involving either:

* High intensity interval training
* Resistance based training (resistance bands will be provided) Researchers will compare the two exercise groups to see if it alters mitochondrial function.

DETAILED DESCRIPTION:
The study will aim to recruit 40 healthy male and female volunteers. They will be assigned into one of three groups;

1. 18 - 35 years old (n=12, 6M:6F)
2. 40 - 55 years old (n=12, 6M:6F)
3. Greater than 65 years old (n=16, 8F:8M)

All volunteers will undergo a full consenting process and undergo a full screening to ensure eligibility prior to commencing the study. If eligible for inclusion in the study, the time commitment will vary from a single half-day study visit, to 12 training sessions over a 4-week period (3 sessions per week) and two half-day study visits (one before and one after the training sessions) depending on the participant's age.

All participants will attend fasted from 22:00 the previous day. Participants will first have a single muscle biopsy of the vastus lateralis before a dual-energy x-ray absorptiometry (DXA) scan to assess body composition and an ultrasound scan of the thigh to assess the muscle structure. A supervised cardiopulmonary exercise testing (CPET) to determine cardiorespiratory fitness will then be performed before a battery of physical function assessments to determine muscle and neuromuscular function. The biopsies will be assessed using an OROBOROS respirometer for the primary endpoint of mitochondrial activity, as well being used to determine cell signaling activity and gene expression.

For those under 65 years of age, a follow-up visit 4-6 days after the biopsy for stitch removal and to complete an end of study questionnaire would be the end of the study. Those volunteers over the age of 65 years will be randomly allocated to a RET group or HIIT group for a 4-week period, after which the assessments from the baseline study day would be repeated. Each exercise group will contain 8 participants (4 male, 4 female).

Training program:

All exercise training will take place within the volunteers own homes in accordance to the divisional policy on this. As well as the education session provided at the baseline study day, participants will be contacted weekly via telephone or video call to encourage participation, to answer any difficulties participants maybe experiencing and to ensure no adverse symptoms are being experienced. A video will be recorded of a member of the research team performing the exercise regimen to enable participants to watch from home.

Each HIIT session last 15 minutes. Participants will be asked to measure their own heart rate during their rest periods and provided with an estimated max heart rate which they should be aiming to achieve within the final 2 exercises. Participants will be provided with a logbook to record the heart rate achieved in each exercise. The regimen will include:

* 2 min warm-up: jogging on the spot
* Each of the following exercises performed for 60seconds, interspaced by 90 seconds rest

  * Star jumps
  * Standing squats
  * On-the-spot sprints
  * Standing squats
  * Star jumps
* 2 min cool-down: jogging on the spot

Each HIIT session lasts an estimated 20minutes. Participants will be provided with a set of TheraBand resistance bands to provide resistance to their workout, and a logbook to record the number of repetitions and band used.

Each session will include:

* 2 min warm-up jogging on the spot
* 2 sets of 12-15 repetitions of:
* Squats
* Hip flexion
* Hip extension
* Hip abduction
* Seated row
* Bench press
* Lateral raises
* 2 min jogging on the spot cooldown.

Each exercise will be separated by 1-minute rest, with participants encouraged to workout to mild fatigue on their final repetition in each set. If able to perform more than the allocated maximum of 15 repetitions prior to fatigue, then participants will be informed to increase the resistance by using a tougher TheraBand.

ELIGIBILITY:
Inclusion Criteria:

* ● Healthy male or female aged over 18 years old able to give informed, written consent.

Exclusion Criteria:

* ● Current participation in a formal exercise regime

  * Inability to use a static exercise bike
  * A BMI <18 or >35 kg/m2
  * Active cardiovascular disease:

    * Uncontrolled hypertension (BP > 160/100)
    * Angina
    * Heart failure (class III/IV)
    * Significant arrhythmia
    * Right to left cardiac shunt
    * Recent cardiac event
  * Taking beta-adrenergic blocking agents
  * Cerebrovascular disease:

    * Previous stroke
    * Aneurysm (large vessel or intracranial)
    * Epilepsy
  * Respiratory disease including:

    * Pulmonary hypertension
    * Significant COPD
    * Uncontrolled asthma
  * Malignancy
  * Clotting dysfunction
  * Significant musculoskeletal or neurological disorders
  * Any suspected or confirmed diagnosis of Covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial activity across age | This will be compared across baseline assessment dates in all ages.
  Mitochondrial oxidative phosphorylation capacity changes seen across the age groups investigated Mitochondrial oxidative phosphorylation capacity will be measured according to oxygen consumption determined by the use of a high-definition respirometer. This will then be compared across ages and expressed as a ratio of maximal consumption.
Mitochondrial activity change with a short-term home-based exercise program in older participants | Assessed prior to and after the completion of a 4 week exercise program
  The effect of either a resistance exercise-based and high-intensity interval training-based home-based training program on mitochondrial function in those over aged 60
  Mitochondrial oxidative phosphorylation capacity will be measured according to oxygen consumption determined by the use of a high-definition respirometer. The changes seen throughout the treatment will then be expressed as a percentage in order to express the changes seen from the baseline.
The altered response to training type | 4 weeks
  The differing responses to either high intensity interval training or resistance based training
  Mitochondrial oxidative phosphorylation capacity will be measured according to oxygen consumption determined by the use of a high-definition respirometer. The changes caused by the training regimen will then be expressed as a percentage in order to express the changes seen from the baseline, and in order to allow comparison between training modality.

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Entry Medical School, University of Nottingham, Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No